CLINICAL TRIAL: NCT02827591
Title: Multimodale Beurteilung Der Stabilität Von Uterusnarbengewebe Bei Z.n. Sectio Caesarea
Brief Title: Assessing the Stability of Uterine Scar Tissue in Women With Previous History of Caesarean Section Using Multimodal Analyses of the Lower Uterine Segment Including Quantitative Sonography
Acronym: QUANTUSLUS
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Gregor Seliger, Dr. med., chief resident, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: QUANTUSLUS
Record Dates: First submitted 2016-07-03; First posted 2016-07-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Scar; Previous Cesarean Section
Keywords: repeat cesarean section; lower uterine segment; quantitative sonography
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Scar tissue is placed in formalin and embedded in paraffin.
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, clinical, observational trial compares the measured value with quantitative ultrasonic (preoperatively) Elastic modulus E (kPA) with the measured value with quantitative ultrasonic Elastic modulus E (kPA) in vitro (postoperatively) and with the experimental measurement done in vitro (postoperatively) of lower uterine segment of women who underwent second cesarean section.

DETAILED DESCRIPTION:
In 1991, 126.297 (15.3%) women delivered by caesarean section in Germany. Since then, the rate of caesarean section increased steadily over the next 20 years, reaching up to 32.2% in 2011. The absolute risk of uterine rupture in vaginal birth after Caesarean section is 1 in 100 deliveries. The risk of perinatal death or the outcome of extremely neurological impairment is 1 in 1000 deliveries.

Statistically more than 300 pregnant women with a prior caesarean delivery visit daily ultrasound departments of german hospitals to investigate the C-section scar before delivery. They have one important question: Is it possible to predict successful trial of labor after cesarean delivery? The information for the risk of uterine rupture remains insufficient based only on ultrasonography assessment.

What are the possibilities of additional parameters to examine the stability of uterine scar tissue? Currently, there is no defined cut-off value of scar thickness for the prediction of uterine rupture. It remains questionable whether the thickness of the lower uterine segment is the determinant factor for the stability of the scar and the probability of rupture. However, another important factor is the functional elasticity or the structure of the connective tissue. It has not been further investigated until now (both quantitatively and qualitatively).

Objective of this project: Multimodalities of assessments, including ultrasonography and elastography, validate the accuracy of uterine scar stability in women with previous history of Caesarean section in vitro and in vivo.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy after previous cesarean section
* pregnancy between 37 0/7 and 42 0/7 weeks of gestation
* primary or secondary indication for cesarean section
* ability to give informed consent in german or english

Exclusion Criteria:

* emergency caesarean section
* <18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pregnancies after previous cesarean section who referre to the tertiary referral care center.
  Pregnant women have been scheduled for a consecutive Caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
In vitro Ultrasonic Elastic Modulus versus in vitro tensile property measurements of LUS | within 1 hour after Cesarean Section
  The measured value of lower uterine segment with quantitative ultrasonic Elastic modulus E (kPA) in vitro versus the experimental tensile property measurements of lower uterine segment done in vitro. (Spearman's rank correlation coefficient)

SECONDARY OUTCOMES:
Difference - In vivo Ultrasonic Elastic Modulus versus in vitro tensile property measurements of LUS | within 1 hour after Cesarean Section
  The measured value of lower uterine segment with quantitative ultrasonic (preoperatively) Elastic modulus E (kPA) in vivo versus the experimental tensile property measurements of lower uterine segment done in vitro (postoperatively). (Spearman's rank correlation coefficient)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Seliger, MD, Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Michael Tchirikov, MD, Study Chair — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varner M. Cesarean scar imaging and prediction of subsequent obstetric complications. Clin Obstet Gynecol. 2012 Dec;55(4):988-96. doi: 10.1097/GRF.0b013e318263c699. PMID 23090468
- [Background] Pollio F, Staibano S, Mascolo M, Salvatore G, Persico F, De Falco M, Di Lieto A. Uterine dehiscence in term pregnant patients with one previous cesarean delivery: growth factor immunoexpression and collagen content in the scarred lower uterine segment. Am J Obstet Gynecol. 2006 Feb;194(2):527-34. doi: 10.1016/j.ajog.2005.07.048. PMID 16458657
- See also: Citations — https://www.aqua-institut.de
- See also: Citations — https://www.destatis.de